CLINICAL TRIAL: NCT02113683
Title: Validation of MMS Test to Detect Active Tumor Growth of Different Cancer Types Before and After Therapy, as Well as for Subsequent Relapse Control in Comparison to Conventional Methods
Brief Title: Validation of MMS Test for Cancer Monitoring
Acronym: MMS-TM
Status: Terminated | Type: Observational
Why Stopped: insufficient recruitment on the part of clinic; study will not resume
Sponsor: MedInnovation GmbH (Industry)
Collaborators: Helios Klinikum Berlin-Buch (Other)
Responsible Party: Sponsor
Other Study IDs: MMS-tm14
Record Dates: First submitted 2014-04-08; First posted 2014-04-15 (Estimated); Last update posted 2018-06-21 (Actual); Status verified 2018-03

CONDITIONS: Colo-rectal Cancer; Stomach Cancer; Melanoma; Sarcoma
Keywords: colo-rectal cancer; stomach cancer; melanoma; MMS test; therapy monitoring; Sarcoma
MeSH Terms: conditions — Colonic Neoplasms; Stomach Neoplasms; Melanoma; Sarcoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- MMS test: therapy monitoring of patients with colo-rectal or stomach disease or with melanoma

SUMMARY:
The purpose of this study is the validation of MMS test to detect active tumor growth in different cancer types before and after therapy, as well as in the course of therapy and for subsequent relapse control compared to standard methods (clinical examination, imaging, tumor markers). It should be consider whether the MMS test has comparable diagnostic accuracy, and thus can replace more expensive or invasive procedures in future.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of colo-rectal cancer
* Clinical diagnosis of stomach cancer
* Suspected diagnosis of melanoma

Exclusion Criteria:

* Colitis ulcerosa
* Morbus Crohn
* Cancer in time period two years before
* Cancer therapy in time period two years before

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with primary diagnosis of cancer
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2014-05; Primary Completion 2018-06-20 (Actual); Study Completion 2018-06-20 (Actual)

PRIMARY OUTCOMES:
active tumor growth before and after cancer therapy | up to 36 month

CONTACTS AND LOCATIONS:
Overall Officials: Katja Waterstradt, PhD, Principal Investigator — MedInnovation GmbH
Locations (1):
- HELIOS Klinikum Berlin-Buch, Klinik für Interdisziplinäre Onkologie, Berlin, Germany